CLINICAL TRIAL: NCT01710345
Title: Safety and Efficacy of Sufentanil NanoTab for Management of Acute Pain Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAP202
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Sufentanil NanoTab 20 mcg (Experimental): Sufentanil NanoTab 20 mcg as needed every 60 minutes for 12 hours
  Interventions: Drug: Sufentanil NanoTab 20 mcg
- Sufentanil NanoTab 30 mcg (Experimental): Sufentanil NanoTab 30 mcg as needed every 60 minutes for 12 hours
  Interventions: Drug: Sufentanil NanoTab 30 mcg
- Placebo NanoTab (Placebo Comparator): Placebo NanoTab as needed every 60 minutes for 12 hours
  Interventions: Drug: Placebo NanoTab

INTERVENTIONS:
Drug: Sufentanil NanoTab 20 mcg
  Arms: Sufentanil NanoTab 20 mcg
Drug: Sufentanil NanoTab 30 mcg
  Arms: Sufentanil NanoTab 30 mcg
Drug: Placebo NanoTab
  Arms: Placebo NanoTab

SUMMARY:
This is a dose-finding study to determine if the sublingual administration of the Sufentanil NanoTab is safe and effective in the treatment of post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for bunion surgery

Exclusion Criteria:

* daily opioid use
* drug or alcohol abuse
* pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lotus Clinical Research, Pasadena, California
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sufentanil NanoTab 20 mcg | Sufentanil NanoTab 30 mcg | Placebo NanoTab
Started | 40 (41 patients were randomized to sufentanil 20 mcg, one patient not dosed due to damaged medication.) | 40 | 20
Completed | 37 | 35 | 19
Not Completed | 3 | 5 | 1
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lack of Efficacy | 2 | 3 | 1
Not completed — Drug Dosing Error | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sufentanil NanoTab 20 mcg | Sufentanil NanoTab 30 mcg | Placebo NanoTab | Total
Number analyzed (Participants) | 40 | 40 | 20 | 100
Age, Categorical [Count of Participants; unit: Participants] — Patients must be at least 18 and no more than 80 years of age
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 39 | 38 | 19 | 96
    >=65 years | 1 | 2 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 10 | 49
  Male | 21 | 20 | 10 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 7 | 12 | 4 | 23
  White | 30 | 26 | 15 | 71
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 4 | 17
  Not Hispanic or Latino | 32 | 35 | 16 | 83
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 20 | 100

OUTCOME MEASURES:

1. Primary Outcome: SPID-12
Description: The primary outcome measure is the summed pain intensity difference over the 12-hour study period (SPID-12). A pain intensity score ranging from 0 (no pain) to 10 (worst possible pain) is obtained at baseline and throughout the 12 hour study period. The SPID-12 is calculated by summing the difference between baseline pain score and pain score at each assessment time point.
  The SPID-12 ranges from -120 (indicative of an increase in pain) to 120 (indicative of a decrease in pain). A higher SPID-12 score is better.
Time Frame: 12 hours
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil NanoTab 20 mcg | Sufentanil NanoTab 30 mcg | Placebo NanoTab
Number analyzed (Participants) | 40 | 40 | 20
units on a scale | -5.65 (2.55) | 6.53 (2.56) | -7.12 (3.64)
Statistical Analysis 1: Comparison: Sufentanil NanoTab 20 mcg vs Placebo NanoTab; Test type: Superiority or Other; p = 0.742, ANCOVA; Mean Difference (Final Values) = 1.47, Standard Error of Mean 4.45
Statistical Analysis 2: Comparison: Sufentanil NanoTab 30 mcg vs Placebo NanoTab; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = 13.66, Standard Error of Mean 4.47

ADVERSE EVENTS:
Time Frame: 12 hours and then time discharge
Arm/Group | Sufentanil NanoTab 20 mcg | Sufentanil NanoTab 30 mcg | Placebo NanoTab
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 23/40 | 30/40 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil NanoTab 20 mcg (N=40) | Sufentanil NanoTab 30 mcg (N=40) | Placebo NanoTab (N=20)
Osteomyeolitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Started 8 days after discharge
Cellulitis (Infections and infestations) | 1 (40) | 0 (0) | 0 (0) — Started 11 days after discharge
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil NanoTab 20 mcg (N=40) | Sufentanil NanoTab 30 mcg (N=40) | Placebo NanoTab (N=20)
Nausea (Gastrointestinal disorders) | 14 | 25 | 0 — AEs occurring at a frequency greater than 5% are included on this list whether or not they were related to study drug
Vomiting (Gastrointestinal disorders) | 11 | 13 | 0
Feeling hot (General disorders) | 3 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 8 | 1
Somnolence (Nervous system disorders) | 2 | 9 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 5 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must be able to review and approve all published